CLINICAL TRIAL: NCT06228742
Title: Molecular Regulation of Skeletal Muscle Anabolic Resistance to Dietary Protein in Response to Injury-mediated Muscle Disuse
Brief Title: Molecular Mechanisms Underlying Anabolic Resistance to Protein Intake During Muscle Disuse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Army Research Institute of Environmental Medicine (U.S. Federal Agency)
Responsible Party: Principal Investigator, Emily E. Howard, Nutrition Physiologist, United States Army Research Institute of Environmental Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 24-02
Record Dates: First submitted 2024-01-18; First posted 2024-01-29 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Atrophy, Disuse; Muscle Atrophy; Muscular Disorders, Atrophic; Disuse Atrophy; Disuse Atrophy Muscle of Thigh
MeSH Terms: conditions — Muscular Disorders, Atrophic; Muscular Atrophy | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Single leg immobilization model consisting of one leg randomly assigned to immobilization with a knee brace and the other leg remaining active and non-immobilized, for 5 days.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immobilized Leg (Experimental): One leg of a young, healthy adult will be randomly assigned to undergo 5 days of immobilization using a rigid knee brace.
  Interventions: Other: Unilateral leg immobilization
- Non-immobilized leg (Experimental): One leg of a young, healthy adult will remain active and not immobilized for 5 days.
  Interventions: Other: Contralateral active leg

INTERVENTIONS:
Other: Unilateral leg immobilization — Participants will have one leg immobilized using a rigid knee brace. Participants will be expected to keep the knee brace on for 5 days and remain non-weight bearing on the immobilized leg. Participants will use crutches to remain non-weight bearing on the immobilized leg.
  Other Names: DISUSE
  Arms: Immobilized Leg
Other: Contralateral active leg — One leg will remain non-immobilized and active during the study. Participants will use this leg to walk with crutches.
  Other Names: ACTIVE
  Arms: Non-immobilized leg

SUMMARY:
This study will characterize intramuscular molecular mechanisms underlying anabolic resistance to protein ingestion during muscle disuse. Adults (n=12) will be studied using a unilateral leg immobilization model in which one leg will be randomly assigned to immobilization and the contralateral, active leg used as a within-subjects control. Immobilization will be implemented for five days using a rigid knee brace, during which time participants will ambulate using crutches. Integrated ribonucleic acid (RNA) synthesis will be determined during immobilization in the immobilized and non-immobilized legs using ingested deuterium oxide, salivary and blood sampling, and muscle biopsies. Immediately after immobilization, muscle biopsies will be collected before and 90 mins after consuming 25 g of whey protein from the immobilized and non-immobilized legs to characterize the intramuscular molecular response to protein feeding. Serial blood samples will be collected during that time to characterize the circulating metabolic response to protein ingestion. Knowledge generated from this effort will inform the development of targeted interventions for mitigating anabolic resistance to protein ingestion that develops during periods of muscle disuse.

DETAILED DESCRIPTION:
Warfighters that sustain musculoskeletal injuries often experience decreased muscle loading and activation post-injury (i.e., muscle disuse) that results in a rapid loss of muscle mass and function. Loss of muscle under these conditions is attributed to a persistent negative net muscle protein balance (muscle protein synthesis [MPS] < muscle protein breakdown [MPB]) that results, in part, from a blunting of MPS in the postprandial state. Nutritional interventions that optimize postprandial MPS have been suggested as countermeasures for this "anabolic resistance" that develops during disuse to preserve muscle mass and accelerate return to duty. However, a poor understanding of mechanisms underlying anabolic resistance during disuse has made it difficult to determine an optimal nutritional intervention. The current study will address this knowledge gap directly by characterizing intramuscular molecular mechanisms underlying anabolic resistance to protein ingestion during muscle disuse. Healthy, recreationally active men and women (n=12) will be studied using a within-subjects, unilateral design. After completing baseline measures of height, weight, and body composition, participants will begin a 3-day run-in phase where they will receive diet instructions (no food provided). Muscle disuse will then be implemented for 5 days using a unilateral leg immobilization model with one leg randomly assigned to immobilization and the contralateral, active leg used as a within-subjects control. Immobilization will be implemented using a rigid knee brace, and participants will ambulate using crutches. Diets will be standardized during the immobilization phase (1.0 g protein/kg/d, 30% of energy intake from fat, and the remaining calories from carbohydrate). Integrated ribonucleic acid (RNA) synthesis will be determined during immobilization in the immobilized and non-immobilized legs using ingested deuterium oxide, salivary and blood sampling, and muscle biopsies. Immediately after immobilization, muscle biopsies will be collected before and 90 mins after consuming 25 g of whey protein from the immobilized and non-immobilized legs to characterize the intramuscular molecular response to protein feeding. Serial blood samples will be collected during that time to characterize the circulating metabolic response to protein ingestion. Knowledge generated from this effort will inform the development of targeted interventions for mitigating anabolic resistance to protein ingestion that develops during periods of muscle disuse.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18-39 years.
* Body mass index (BMI) between 18.5-30 kg/m2
* Healthy without evidence of chronic illness (e.g., diabetes, cardiovascular disease, Crohn's disease) or musculoskeletal injury as determined by the USARIEM Office of Medical Oversight (OMSO) or home duty station medical support.
* Routinely participate in aerobic and/or resistance exercise at least 2 days per week.
* Willing to refrain from alcohol, smoking, smokeless nicotine products (includes e-cigarettes, vaping, chewing tobacco), caffeine, and dietary supplements (i.e., vitamin D, probiotics) during the run-in diet, immobilization phase, and final testing day of the study.
* Supervisor approval for federal civilian employees and non-human research volunteer (HRV) active-duty military personnel stationed at Natick Soldier System Center (NSSC).
* Biological females must have normal menstrual cycles between 26-32 days in duration; 5 menstrual cycles within the past 6 months; or on continuous hormonal contraception (i.e., intrauteraine device (IUD) or oral contraceptives without placebo).

Exclusion Criteria:

* Musculoskeletal injuries that may interfere with the safe use of crutches.
* Personal or family history of thrombosis, or prior diagnosis of deep vein thrombosis (DVT) or pulmonary embolism (PE).
* Metabolic or cardiovascular abnormalities, gastrointestinal disorders, neuromuscular disorders, lower-limb amputation, or muscle/bone wasting disorders (e.g., diabetes, cardiovascular disease, Crohn's disease, etc.).
* Significantly abnormal blood clotting as determined by OMSO or home duty station medical support.
* Allergy to lidocaine (or similar local anesthetic)
* Present condition of alcoholism, anabolic steroid use, or other substance abuse issues as determined by OMSO or home duty station medical support.
* Blood donation within 8-wk of beginning the study.
* Pregnant, trying to become pregnant, and/or breastfeeding (results of urine pregnancy test and self-report for breastfeeding will be obtained before body composition testing).
* Unwilling or unable to consume study diets or foods provided due to personal preference and/or food allergies.
* Unwilling or unable to adhere to study physical restrictions (i.e., no structured physical activity or recreational activity beyond activities of daily living) 24 hours before and during immobilization, and the final testing day.
* Unwilling or unable to keep the knee brace on and walk with crutches during the immobilization phase.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2024-02-20 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Integrated ribonucleic acid (RNA) synthesis | 5 days
  deuterium oxide coupled with muscle biopsies
Intramuscular protein signaling response to protein ingestion | 90 minutes
  muscle biopsies to assess protein signaling response to consuming 25 g of whey protein

CONTACTS AND LOCATIONS:
Overall Officials: Emily E Howard, PhD, Principal Investigator — US Army Research Institute of Environmental Medicine
Locations (1):
- US Army Research Institute of Environmental Medicine, Natick, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No